CLINICAL TRIAL: NCT02983318
Title: Molecular Imaging of Brain Inflammation in Depressive Disorders
Acronym: DiME
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 100128
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder, Major; Positron-Emission Tomography
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood drawn and analyzed
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/MRI using 18[F]EPPA ligand: given experimental ligand FEPPA during MRI/PET scan to identify glutamate activity in the brain using FEPPA ligand

SUMMARY:
In a number of neuropsychiatric disorders such as depression, both brain inflammation and glutamate mediated excitotoxicity (cell death through over-activated stimulation) are suspected to play a key role. It is difficult, if not impossible, to determine the potential destructiveness of the inflammatory response seen in disease states by studying the brain's inflammatory cells (microglia) activity in isolation. The investigators are proposing to develop the means to concurrently study inflammatory response (i.e., microglial activity) and its potentially devastating consequence (i.e., glutamate excitotoxicity) across the entire brain in order to establish the importance of inflammation. In this study the investigators propose a phased clinical study whereby the early-phase involves the development of our capacity to study inflammation-mediated damage to brain cells, followed by a feasibility study in patients with clinical depression that tests whether concurrent inflammation and glutamate excess could be measured in key brain regions associated with a depressed mood state.

ELIGIBILITY:
Inclusion Criteria:

* screening form for MRI/PET is satisfactory after being reviewed by a radiologist
* diagnosed with depression or healthy control participants with no present mental health disorder
* Good general health with no diseases expected to interfere with the study
* Subject is not pregnant, lactating, or of childbearing potential (must be practicing effective form of birth control)
* Patient and healthy controls must not have an infection or an autoimmune disorder or persistent inflammation.

Exclusion Criteria:

* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* use of Investigational agents within last month

Ages: 19 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Able to pass MRI screening form (reviewed by a MRI technician)
  * diagnosed with depression or healthy control participants with no present mental health disorder
  * Good general health with no diseases expected to interfere with the study
  * Subject is not pregnant, lactating, or of childbearing potential (must be practising effective form of birth control)
  * Patient and healthy controls must not have an infection or an autoimmune disorder or persistent inflammation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
inflammation-related excitotoxicity in the brain | single time. Data collected at baseline with no follow up.
  Cross sectional MRI/PET scan will be used to identify inflammation related excitotoxicity in the brain in healthy individuals and those diagnosed with major depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Palaniyappan, MBBS/PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No